CLINICAL TRIAL: NCT03288402
Title: Investigation of the Effects of Breakfast or Caffeine Containing Beverages on the Measurement of Plasma Chromogranin A in Patients With Gastro-entero-pancreatic Neuroendocrine Tumours (GEP-NET)
Brief Title: Investigation of the Effects of Diet on the Measurement of Plasma Chromogranin in NET Patients
Acronym: DIB-NET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: MW165915/IRAS ID 197653
Record Dates: First submitted 2017-08-10; First posted 2017-09-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Intervention Model Description: double crossover (ongoing fasted; or caffeine containing beverages; of 5-item English breakfast)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ongoing fasted (Experimental): ongoing fasted following 10 h overnight fast; series blood samples CgA over 180 min
  Interventions: Other: ongoing fasted state, intake of caffeine containing beverages or 5-item English breakfast
- intake of caffeine containing beverages (Experimental): 10 h overnight fast; intake of caffeine containing beverages; series blood samples CgA over 180 min
  Interventions: Other: ongoing fasted state, intake of caffeine containing beverages or 5-item English breakfast
- intake of 5 item English breakfast (Experimental): 10 h overnight fast; intake of 5-item English breakfast; series blood samples CgA over 180 min
  Interventions: Other: ongoing fasted state, intake of caffeine containing beverages or 5-item English breakfast

INTERVENTIONS:
Other: ongoing fasted state, intake of caffeine containing beverages or 5-item English breakfast — effects of ongoing fasted state; or intake caffeine containing beverages; or 5-item English breakfast on plasma CgA measurements, in series blood tests every 30 min over 180 min

SUMMARY:
Measurement of plasma chromogranin A remains the most commonly used biomarkers for both screening and monitoring of patients with gastro-entero-pancreatic neuroendocrine tumours (GEP-NET), despite several limitations that include: lack of a reference CgA standard; wide variations depending on the used assay in different laboratories; and varying sensitivity ranges from 60 to 90% with low specificity <50%, depending on the population studied.

Surprisingly, and to the best of our knowledge, only three studies with small numbers of participants have been published that have investigated possible effects of food intake on the measurement of CgA. Most have been performed in healthy controls or patients on treatment with proton pump inhibitors for chronic gastritis (up to n = 11 per group) but only one study has investigated patients with GEP-NET, where n = 6 patients with gastric NET were included.

In this study, the investigators aim to assess the time dependent effects of normally ingested diet (5-item English breakfast; or tea or coffee; or ongoing fasted state) on plasma chromogranin A measurements, using timed measurements over 180 min following an > 10 hours overnight fast, in a randomised double-crossover design. The investigators aimed to include 25 - 35 patients with a histologically confirmed diagnosis of a GEP-NET of varying primary tumour location, tumour stage, grade; and presence or absence of treatment with long acting somatostatin analogues; as well as 10 - 15 healthy controls. In an additional small subgroup of patients who are initiated on treatment with GLP-1 analogues i.e. for type 2 diabetes or obesity, the investigators aim to establish whether injection of GLP-1 analogues has any effects on plasma CgA measurements.

ELIGIBILITY:
Inclusion Criteria:

GEP-NET patients:

* Confirmed diagnosis of NET
* Aged 18 or over
* Able to provide written informed consent
* Able to commit to 3 visits within a 4 week period
* Able to fast overnight
* Able to adequately read/write/speak English

CONTROLS:

* No known diagnosis of NET
* Aged 18 or over
* Able to provide written informed consent
* Able to commit to 3 visits within a 4 week period
* Able to fast overnight
* Able to adequately read/write/speak English

Exclusion Criteria:

- GEP-NET patients

* No confirmed diagnosis of a NET
* Under the age of 18
* Unable to provide written informed consent
* Pregnant women
* Any patients who are un well on the day of their routine appointment
* Unable to fast overnight
* Unable to adequately read/write/speak English

CONTROLS

* Confirmed diagnosis of NET
* Under the age of 18
* Unable to provide written informed consent
* Pregnant women
* Any patients who are un well on the day
* Unable to fast overnight
* Unable to adequately read/write/speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
changes in plasma CgA measurements related to intake of food or caffeine containing beverages, as compared to ongoing fasted state | up to 180 min
  plasma CgA 0, 30, 60, 90, 120, 150 and 180 min

CONTACTS AND LOCATIONS:
Overall Officials: Martin O Weickert, Professor, Study Chair — The ARDEN NET Centre, ENETS CoE; Megan Symington, Dr, Principal Investigator — The ARDEN NET Centre, ENETS CoE; Helen Robbins, Dr, Principal Investigator — The ARDEN NET Centre, ENETS CoE
Locations (1):
- The ARDEN NET Centre, ENETS Centre of Excellence, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: publication list MO Weickert — https://www.ncbi.nlm.nih.gov/pubmed/?term=weickert+mo